CLINICAL TRIAL: NCT07214584
Title: Using Plasma Human Papillomavirus (HPV)-Related Deoxyribonucleic Acid (DNA) and Ribonucleic Acid (RNA) to Follow Response of Cervical Cancer to Surgery, Radiation, and Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRB202501136
Record Dates: First submitted 2025-10-07; First posted 2025-10-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer; Human Papilloma Virus (HPV)
Keywords: HPV; HPV Positive Cervical Cancer; Cervical Cancer; Recurrent Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual whole blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to test two commercially available technologies for their ability to detect treatment response in patients with cervical cancer following surgery, radiation, and chemotherapy: one based on polymerase chain reaction (PCR; NavDx) and the other on branched DNA (Quantivirus HPV [DNA]). A 9-month feasibility study will be performed to examine the side-by-side utility of both NavDx and Quantivirus HPV DNA assays in predicting cervical cancer treatment response.

These tests could prove to be highly sensitive methods for evaluating minimal residual disease and for quantitation of response to surgery, radiation, and chemotherapy in patients with cervical cancer.

Primary Goal:

Feasibility for NavDx HPV DNA assay (Naveris, Inc) to be used for personalized prediction of tumor response before and after treatment.

Secondary Goals:

1. Comparability of the Quantivirus HPV DNA/mRNA assay (DiaCarta, Inc) with the NavDx HPV DNA assay and,
2. Feasibility of the Quantivirus technology for measuring treatment response within the first day to 2 weeks of radiation, surgery, or a new chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* HPV-associated squamous cell, adenocarcinoma, or adenosquamous cancers of the uterine cervix with evaluable disease
* Diagnosed with American Joint Committee on Cancer (AJCC) stage I or higher, or metastatic disease.
* Presence of evaluable disease on pre-treatment standard of care imaging with plans to obtain serial post-treatment standard of care imaging
* Agree to perform the required research-related blood tests and cervical mucous testing.

Exclusion Criteria:

* Unable to consent or refusal to sign a consent form
* Not meet any inclusion criteria
* Unable to comply with follow up scheduling.
* Diagnosed with a synchronous malignancy requiring cancer-directed therapy

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients with HPV associated cancers of the uterine cervix with active, evaluable/measurable disease.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Circulating HPV DNA/mRNA Liquid Biopsy for Evaluating Treatment Response in Cervical Cancer | From enrollment to the end of the first surveillance visit, which occurs at 3-4 months post op or post-chemo, or at the patient's 3-4 month follow-up radiation therapy visit.
  This is a feasibility study to determine the sensitivity of circulating HPV DNA/mRNA, measured by either or both NavDx or Quantivirus as a liquid biopsy, to evaluate treatment response in cervical cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No